CLINICAL TRIAL: NCT01303185
Title: Pulsed Dye Laser for the Psoriatic Nail
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ying-Yi Chiang, Attending Physician, Taipei Medical University WanFang Hospital
Other Study IDs: 99074
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Psoriatic Nail
Keywords: Psoriatic Nail; Pulsed dye laser

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
The treatment options for nail psoriasis have been limited, and the management of nail psoriasis has been challenging for physicians.To evaluate the effect of pulsed dye laser (PDL) in the treatment of nail psoriasis.

DETAILED DESCRIPTION:
Psoriatic nails of patient's right hand were treated using PDL (595 nm) .The pulsed duration is 1.5ms, the beam diameter is 7mm, and the laser energy is 8.0 to 10.0 J/cm2. The treatment course of pulse dye laser is once monthly for 6 months. Psoriatic nails of both hands are treated with Tazarotene cream for 6 months. Clinical efficacy is statistically evaluated according to Nail Psoriasis Severity Index (NAPSI) score differences between right and left hand one month after 3rd and 6th therapy.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic nail refractory to other topical and systemic treatment therapy
* ≧ 16 years old

Exclusion Criteria:

* Patient with pregnancy
* Patient with photo sensitivity
* Patient with severe wound around finger nails or paronychia
* Patient with hypersensitivity to Tazarotene cream

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Psoriatic nail patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
NAPSI | 3rd and 6th months
global physician assessment | 3rd and 6th months

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Yi Chiang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan